CLINICAL TRIAL: NCT00240435
Title: A Randomized, Double-blind, Double-dummy, Placebo- and Active-controlled, Parallel Group Efficacy and Safety Comparison of 12-week Treatment of Two Doses (5 Mcg and 10 Mcg) of Tiotropium Inhalation Solution Delivered by the Respimat Inhaler, Placebo and Ipratropium Bromide Inhalation Aerosol (MDI) i
Brief Title: 12 Week Comparison of 5 Mcg and 10 Mcg of Tiotropium / Respimat, Placebo and Ipratropium MDI in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.252
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Device: 5 mcg once daily tiotropium inhalation solution delivered by the Respimat inhaler
Device: 10 mcg once daily tiotropium inhalation solution delivered by the Respimat inhaler

SUMMARY:
The primary objective was to compare the bronchodilator efficacy of two doses (5 mcg and 10 mcg) of tiotropium inhalation solution delivered by the Respimat inhaler once daily to placebo and to ipratropium bromide MDI four times daily in patients with COPD. The secondary objective was to compare the safety of tiotropium inhalation solution delivered by the Respimat to placebo and ipratropium bromide MDI.

ELIGIBILITY:
Outpatients of either sex, aged >/= 40 years with a diagnosis of COPD (FEV1 </= 60% predicted [ECCS criteria] and FEV1/FVC </= 70%)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491
Dates: Start 2002-11; Primary Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Trough FEV1 response after 12 weeks of treatment. | after 12 weeks

SECONDARY OUTCOMES:
Trough FEV1 response | after 1, 4 and 8 weeks
Trough FVC response | after 1, 4, 8 and 12 weeks
FEV1 and FVC area under the curve and peak response | after 0, 1, 4, 8 and 12 weeks
Individual FEV1 and FVC measurements at each time point | during study course of 12 weeks
Therapeutic response and percentage of responders | after 0 and 12 weeks
Weekly mean pre-dose morning and evening PEFR | during study course of 12 weeks
Number of occasions of rescue therapy used per day (PRN salbutamol) | during study course of 12 weeks
COPD symptom scores | during 15 weeks
Physician's Global Evaluation | during 15 weeks
Number of patients with at least one exacerbation of COPD | 15 weeks
time to first exacerbation | 15 weeks
number of exacerbations | 15 weeks
number of exacerbation days | 15 weeks
Patient satisfaction and preference | 12 weeks
All adverse events | during 15 weeks, follow-up period included
Pulse rate and blood pressure for the first three hours following dosing | after 0, 1, 4, 8 and 12 weeks
Routine blood chemistry, haematology and urinalysis | after 12 weeks
12-lead ECG | after 12 weeks
Physical examination | after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (25):
- United States (14):
  - Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, Downey, California
  - University of California - Los Angeles, Los Angeles, California
  - Boehringer Ingelheim Investigational Site, Palo Alto, California
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Boehringer Ingelheim Investigational Site, Bay Pines, Florida
  - Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - Boehringer Ingelheim Investigational Site, Wheaton, Maryland
  - Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - Boehringer Ingelheim Investigational Site, Elizabeth City, North Carolina
  - Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - Boehringer Ingelheim Investigational Site, Dallas, Texas
- Canada (11):
  - Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Boehringer Ingelheim Investigational Site, Courtice, Ontario
  - St. Joseph's Hospital Cardiac Research, Hamilton, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Department of Respiratory Medicine, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - SMBD--Jewish General Hospital, Montreal, Quebec
  - Centre de Recherche Clinique -CUSE, Sherbrooke, Quebec
  - Hopital Laval, Ste-Foy, Quebec
  - c/o Hemodynamics Offices, Saskatoon, Saskatchewan